CLINICAL TRIAL: NCT04002310
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Intravitreal Doses and Multiple Intravitreal Dosing of BI 754132 in Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration (Open Label, Non-randomized, Uncontrolled).
Brief Title: A Study to Test How Well Different Doses of BI 754132 Are Tolerated in Patients With an Advanced Form of Age-related Macular Degeneration Called Geographic Atrophy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was discontinued in the interests of patients considering benefit/risk balance.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1418-0001; 2018-004125-92 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 0.3 mg BI 754132 - SRD part (Experimental): 0.3 milligram (mg) BI 754132 powder for solution for injection 60mg/vial with solution of diluent was administered intravitreally as one single injection on Day 1. One patient was dosed first, and when the safety assessments through Day 4 showed no ophthalmological dose limiting events (DLEs) or systemic DLEs, the remaining patients were dosed. Single rising dose (SRD) part.
  Interventions: Drug: BI 754132
- 1 mg BI 754132 - SRD part (Experimental): 1 mg BI 754132 powder for solution for injection 60mg/vial with solution of diluent was administered intravitreally as one single injection on Day 1. One patient was dosed first, and when the safety assessments through Day 4 showed no ophthalmological dose limiting events (DLEs) or systemic DLEs, the remaining patients were dosed. SRD part.
  Interventions: Drug: BI 754132
- 3 mg BI 754132 - SRD part (Experimental): 3 mg BI 754132 powder for solution for injection 60mg/vial with solution of diluent was administered intravitreally as one single injection on Day 1. One patient was dosed first, and when the safety assessments through Day 4 showed no ophthalmological dose limiting events (DLEs) or systemic DLEs, the remaining patients were dosed. SRD part.
  Interventions: Drug: BI 754132
- 6 mg BI 754132 - SRD part (Experimental): 6 mg BI 754132 powder for solution for injection 60mg/vial with solution of diluent was administered intravitreally as one single injection on Day 1. One patient was dosed first, and when the safety assessments through Day 4 showed no ophthalmological dose limiting events (DLEs) or systemic DLEs, the remaining patients were dosed. SRD part.
  Interventions: Drug: BI 754132
- 6 mg BI 754132 - MD part (Experimental): 6 mg BI 754132 powder for solution for injection 60mg/vial with solution of diluent was administered intravitreally as 3 injections, each separated by 4 weeks (that is, Day 1, Day 29 and Day 57). Multiple dose.
  Interventions: Drug: BI 754132

INTERVENTIONS:
Drug: BI 754132 — One single injection

SUMMARY:
This is a study in adults with geographic atrophy, an advanced form of age-related macular degeneration. The purpose of this study is to find out how well different doses of BI 754132 are tolerated.

The participants are in the study for about 4 months. During this time, they visit the study site about 10 times. Participants receive 1 injection of BI 754132 directly into one of the eyes affected by geographic atrophy. In this study, BI 754132 is given to humans for the first time.

The doctors compare how well participants tolerate the different doses of BI 754132. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion criteria:

- Men and women with Geographic Atrophy (GA) secondary to Age-related Macular Degeneration (AMD): For the SRD part, the GA lesion in the study eye must be ≥ 1.9 mm2 disc area in size (approximately ≥ 0.75 disc area in size); For the MD part the total GA lesion size in the study eye must be ≥ 7.5 mm2 (approximately ≥ 3 disc area in size)

* Fellow eye is not required to have GA
* Best Corrected Visual Acuity (BCVA):

  * SRD part: BCVA of 20/100 to 20/400 Snellen (corresponding to 19 to 53 letters in the ETDRS chart) in the study eye equivalent measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol
  * MD part: BCVA score of ≤53 letters (Snellen equivalent of 20/100) in the study eye
* Age ≥ than 50 years
* Best-corrected VA in the non-study eye must have a better best-corrected VA compared to the study-eye
* Women of childbearing potential (WOCBP) cannot be included. Men able to father a child must be ready and able to use highly effective methods of birth control per International Council on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed informed consent consistent with International Council on Harmonisation Good Clinical Practice (ICH GCP) guidelines and local legislation prior to participation in the trial, which includes medication washout and restrictions
* Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order

Exclusion criteria

* GA in either eye because of causes other than AMD
* History of choroidal neovascularization (CNV) in the study eye and in the fellow eye
* Previous treatment in the study eye for GA secondary to AMD within 6 months prior to screening visit (ongoing therapy with vitamin and mineral supplements is allowed)
* Additional eye disease in the study eye that could compromise

  * best corrected VA (BCVA) with visual field loss,
  * uncontrolled glaucoma intraocular pressure (IOP>24),
  * clinically significant diabetic maculopathy,
  * history of ischemic optic neuropathy or retinal vascular occlusion,
  * symptomatic vitreomacular traction,
  * genetic disorders such as retinitis pigmentosa);
  * history of high myopia > 8 diopters in the study eye and
  * anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with Spectral Domain Optical Coherence Tomography (SD-OCT)
* Any prior intraocular surgery in the study eye other then uneventful lens replacement for cataract within 3 months prior to screening
* Aphakia or total absence of the posterior capsule. Yttrium aluminum garnet (YAG) laser capsulotomy permitted, more than 3 month prior to enrollment in the study eye
* Current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol)
* Significant disease or other medical conditions (as determined by medical history, examination and clinical investigations at screening) that may, in the opinion of the investigator result in the any of the following:

  * Put the patient at risk because of participation in the study
  * Influence the results of the study,
  * Cause concern regarding the patient's ability to participate in the study, e.g. cardiac (including tachycardia), gastro-intestinal, hepatic, renal, metabolic, dermatologic, neurological, haematological, oncological and psychiatric.
* Patients with malignancy for which the patient has undergone resection, radiation or chemotherapy within past 5 years. Patients with treated basal cell carcinoma or fully cured squamous cell carcinoma are allowed.
* Known hypersensitivity to any of the ingredients used in the Investigational Medical Product (IMP) formulation, or any of the medications used
* Active intraocular inflammation in the study eye
* Active infectious conjunctivitis in either eye
* Further exclusion criteria apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Specialty Institute, Pensacola, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
- United Kingdom (5):
  - Bristol Eye Hospital, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open label, non-randomized, uncontrolled trial to test how single rising intravitreal doses and multiple doses of BI 754132 are tolerated in patients with geographic atrophy. Recruitment was to be done successively for the dose groups. The multiple dose (MD) part recruited patients only after the single rising dose (SRD) part was completed and safety of the selected dose was endorsed by the safety monitoring committee.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 6 mg BI 754132 - MD Part: 6 mg BI 754132 powder for solution for injection 60mg/vial with solution of diluent was administered intravitreally as 3 injections, each separated by 4 weeks (that is, Day 1, Day 29 and Day 57). Multiple dose (MD) part.
Period: Overall Study
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part | 6 mg BI 754132 - MD Part
Started | 3 | 3 | 3 | 6 | 3
Treated | 3 | 3 | 3 | 6 | 3
Completed (Completed=Not prematurely discontinued from trial medication.) | 3 | 3 | 3 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor put on hold on treatment plan. | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS consisted of all patients who were treated with at least 1 dose of BI 754132.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part | 6 mg BI 754132 - MD Part | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.3 (4.9) | 78.7 (2.5) | 70.7 (8.1) | 77.7 (6.0) | 77.3 (8.3) | 76.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5 | 2 | 12
  Male | 1 | 2 | 1 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 6 | 3 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SRD Part: Number of Patients With Ocular (in the Study Eye) or Systemic Dose Limiting Events (DLEs)
Description: SRD part: Number of patients with ocular or systemic DLEs from drug administration. Systemic DLEs were defined as drug-related adverse events (AEs), as defined by the investigator, of moderate or severe intensity on the Common terminology criteria for adverse events (CTCAE) scale, and included diarrhea, cough, or patient-reported paraesthesia, dysgeusia, taste abnormality, taste disorder, or hyposmia. Single rising dose (SRD) part.
Time Frame: From drug administration until end of trial, up to 100 days.
Population: Treated Set (TS): The TS consisted of all patients who were treated with at least 1 dose of BI 754132. Only participants included in the SRD part.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: MD Part: Number of Patients With Drug Related Adverse Events (AEs)
Description: Number of patients with drug-related adverse events (AEs). Multiple dose (MD) part.
Time Frame: From drug administration until end of trial, up to 155 days
Population: Treated Set (TS): The TS consisted of all patients who were treated with at least 1 dose of BI 754132. Only participants included in the MD part.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg BI 754132 - MD Part
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: SRD Part: Number of Patients With Drug-related Adverse Events (AEs)
Description: Number of patients with drug-related AEs. Single rising dose (SRD) part.
Time Frame: From drug administration until end of trial, up to 100 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 1 | 0 | 1 | 1

4. Secondary Outcome: SRD Part: Number of Patients With Any Ocular Adverse Events (AEs) in the Study Eye
Description: Number of patients with any ocular adverse events in the study eye. Single rising dose (SRD) part.
Time Frame: From drug administration until end of trial, up to 100 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 1 | 1 | 2 | 2

5. Secondary Outcome: SRD Part: Maximum Serum Concentration of BI 754132 After a Single Intravitreal Dose (Cmax)
Description: Maximum serum concentration of BI 754132 after a single intravitreal dose (Cmax). Single rising dose (SRD) part.
Time Frame: At Day 1, 4, 8, 15, 29, 56, 84 and Day 100.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all patients in the treated set (TS) who provided at least 1 plasma sample for determination of PK parameters and whose data were not excluded due to a protocol violation relevant to the evaluation of the PK or due to PK non-evaluability. Only SRD part. For the 6 mg arm: Only patients with measurable serum concentration of BI (2 out of 6) are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 2
nanogram/milliliter (ng/mL) | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | 26.9 (2.55)

6. Secondary Outcome: SRD Part: Area Under the Concentration-time Curve of BI 754132 in Serum Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 754132 in serum over the time interval from 0 extrapolated to infinity (AUC0-∞). Singe rising dose (SRD) part.
Time Frame: At Day 1, 4, 8, 15, 29, 56, 84 and Day 100.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter (h*ng/mL)
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 2
Hours*nanogram per milliliter (h*ng/mL) | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | 4620 (2220)

7. Secondary Outcome: SRD Part: Time From Dosing to Maximum Serum Concentration of BI 754132 (Tmax)
Description: Time from dosing to maximum serum concentration of BI 754132 (tmax). Single rising dose (SRD part).
Time Frame: At Day 1, 4, 8, 15, 29, 56, 84 and Day 100.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours (h)
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 2
Hours (h) | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | NA (NA) — Results could not be calculated, as none of the patients had sufficient measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132. | 72.5 (96.9)

8. Secondary Outcome: MD Part: Trough Levels of BI 754132 Before Second Administration (Cmin,1)
Description: Systematic exposure of BI 754132 after multiple intravitreal doses as assessed by Cmin,1 (trough levels of BI 754132 before second administration). Multiple dose (MD) part.
Time Frame: Up to 29 days.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all patients in the treated set (TS) who provided at least 1 plasma sample for determination of PK parameters and whose data were not excluded due to a protocol violation relevant to the evaluation of the PK or due to PK non-evaluability. Only MD part.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | 6 mg BI 754132 - MD Part
Number analyzed (Participants) | 3
Nanogram/milliliter (ng/mL) | NA (NA) — Not calculable, as none of the patients had any measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132.

9. Secondary Outcome: MD Part: Trough Levels of BI 754132 Before Third Administration (Cmin,2)
Description: Systematic exposure of BI 754132 after multiple intravitreal doses as assessed by Cmin,2 (trough levels of BI 754132 before third administration). Multiple dose (MD) part.
Time Frame: Up to 57 days.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | 6 mg BI 754132 - MD Part
Number analyzed (Participants) | 3
Nanogram/milliliter (ng/mL) | NA (NA) — Not calculable, as none of the patients had any measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132.

10. Secondary Outcome: MD Part: Plasma Concentration of BI 754132 4, 8 and 14 Weeks After the Third Administration
Description: Plasma concentration of BI 754132 4, 8 and 14 weeks after the third administration. Multiple dose (MD) part.
Time Frame: At Day 85, 113 and Day 155.
Population: as for outcome 8
Measure: Number; unit: Nanogram/milliliter (ng/mL)
Arm/Group | 6 mg BI 754132 - MD Part
Number analyzed (Participants) | 3
Nanogram/milliliter (ng/mL)
  4 weeks after the third administration | NA — Not calculable, as none of the patients had any measurable (i.e. above lower limit of quantification (LLOQ)) serum concentration of BI 754132.
  8 weeks after the third administration | NA — Not calculable, as none of the patients had any measurable (i.e. above LLOQ) serum concentration of BI 754132.
  14 weeks after the third administration | NA — Not calculable, as none of the patients had any measurable (i.e. above LLOQ) serum concentration of BI 754132.

ADVERSE EVENTS:
Time Frame: From first drug administration until end of trial, up to 100 days for single rising dose (SRD) part and up to 155 days for multiple dose (MD) part. For BI 754132, the residual effect period (REP) after Intravitreal (IVT) administration is not known. Therefore, all adverse events with an onset between start of treatment and end of trial (EOT) visit were assigned to the on-treatment period.
Description: Treated Set (TS): The TS consisted of all patients who were treated with at least 1 dose of BI 754132.
Arm/Group | 0.3 mg BI 754132 - SRD Part | 1 mg BI 754132 - SRD Part | 3 mg BI 754132 - SRD Part | 6 mg BI 754132 - SRD Part | 6 mg BI 754132 - MD Part
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/6 | 2/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 3/3 | 3/6 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg BI 754132 - SRD Part (N=3) | 1 mg BI 754132 - SRD Part (N=3) | 3 mg BI 754132 - SRD Part (N=3) | 6 mg BI 754132 - SRD Part (N=6) | 6 mg BI 754132 - MD Part (N=3)
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 1 | 1
Papilloedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg BI 754132 - SRD Part (N=3) | 1 mg BI 754132 - SRD Part (N=3) | 3 mg BI 754132 - SRD Part (N=3) | 6 mg BI 754132 - SRD Part (N=6) | 6 mg BI 754132 - MD Part (N=3)
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vitreous opacities (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated prematurely based on a negative benefit-risk assessment, which was based on the analysis of the safety data during the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04002310/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT04002310/SAP_001.pdf